CLINICAL TRIAL: NCT02589899
Title: Monitoring of Needle-placement With Multiple Frequency Bioimpedance Monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Axel Rudolf Sauter, PhD, Oslo University Hospital
Other Study IDs: impedance monitoring 1/2015
Record Dates: First submitted 2015-10-22; First posted 2015-10-28 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Electric Impedance; Human; Hypodermic Needles; Tissues; Nerve

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Needle placement in different tissue types: Needle placement and impedance measurements in different tissue types
  Interventions: Other: Needle placement in different tissue types

INTERVENTIONS:
Other: Needle placement in different tissue types — Bioimpedance will be measured for needle positions in different tissue types

SUMMARY:
A novel algorithm for bioimpedance measurements to detect nerve tissue, and discriminate it from other tissue types has been developed in a porcine model, by analysing a complex impedance dataset based on multiple measurement frequencies. It must now be confirm that the previous results are applicable in humans. Measurements from 24 predefined needle positions will be obtained in 16 of the 32 volunteers that are included in the study (part A). A new algorithm to detect nerve tissue will be developed based on these measurement results. Further impedance algorithms will be developed for other tissue type. The efficacy of the algorithms (sensitivity and specificity) will be evaluated in the 16 following volunteers (part B).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* American society of anaesthesiologists score (ASA) 1 or 2
* Volunteers that have given informed written consent

Exclusion Criteria:

* Volunteers that cannot cooperate for the examination
* Volunteers with neurologic disease, nerve- or vascular impairment
* ASA > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Success in the identification of nerve tissue by the use of an algorithm based on a multiple frequency impedance measurement (MFIM) algorithm. The outcome is binary (success vs failure). | From day 1 up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Kalvoy H, Sauter AR. Detection of intraneural needle-placement with multiple frequency bioimpedance monitoring: a novel method. J Clin Monit Comput. 2016 Apr;30(2):185-92. doi: 10.1007/s10877-015-9698-3. Epub 2015 Apr 23. PMID 25902898